CLINICAL TRIAL: NCT02846948
Title: The Impact of Extended Hemodynamic Monitoring by Focused Transthoracic Echocardiography in Urgent Abdominal Surgery for Septic Patients
Brief Title: The Impact of Focused Transthoracic Echocardiography in Urgent Abdominal Surgery for Septic Patients
Acronym: ECHOCARD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lithuanian University of Health Sciences (Other)
Responsible Party: Principal Investigator, Asta Maculiene, Principal Investigator, Lithuanian University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MIP051/2015
Record Dates: First submitted 2016-07-25; First posted 2016-07-27 (Estimated); Last update posted 2018-11-21 (Actual); Status verified 2018-11

CONDITIONS: Sepsis; Hypovolemia; Peritonitis
Keywords: sepsis; echocardiography; urgent; abdominal surgery
MeSH Terms: conditions — Sepsis; Hypovolemia; Peritonitis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Non-echo group (No Intervention): Patients get the standard monitoring and treatment based on Good medical practice. Extended monitoring by focused echocardiography is not applied for this group.
- Focussed echocardiography group (Experimental): The extended cardiac monitoring by focused assessed transthoracic echocardiography is applied.
  Interventions: Other: Focused assessed echocardiography

INTERVENTIONS:
Other: Focused assessed echocardiography — Focused assessed transthoracic echocardiography is non-invasive, painless procedure. The transducer is placed on the chest at certain locations and angles to get the required information on patient's condition.
  Arms: Focussed echocardiography group

SUMMARY:
The aim of the study is to identify the diagnostic value of the focused assessed echocardiography in septic patients undergoing urgent abdominal surgery due to peritonitis. The investigators expect that the incidence of hemodynamic instability will be reduced and the survival of the patients will be improved.

DETAILED DESCRIPTION:
Often sepsis remains undiagnosed at the very beginning because of the concentration to the surgical pathology in perioperative period. This results in unacceptably high mortality. The investigators hypothesize that extended hemodynamic monitoring by focused transthoracic echocardiography will personalize early fluid resuscitation which will improve patient's outcome.

The goals of the investigators study are:

* To conduct two-group randomized controlled clinical trial to compare patient management based on standard monitoring and extended hemodynamic monitoring by focused transthoracic echocardiography in patients undergoing urgent abdominal surgery due to peritonitis.
* To demonstrate that patient management based on extended hemodynamic monitoring by focused echocardiography results in improved survival, reduced incidence of hemodynamic instability during perioperative period.
* To compare an amount of administrated of intravenous fluids in both groups.

The investigators hypothesize that focused echocardiography monitoring will result in more administrated intravenous fluids during perioperative period.

ELIGIBILITY:
Inclusion Criteria:

* Age more than 18 years old.
* Patients undergoing urgent abdominal surgery due to diffuse peritonitis.
* SOFA score >2.
* Patients who sign an agreement to participate in the study.

Exclusion Criteria:

* Younger than 18 years old.
* Known pregnancy.
* Unconscious patients or those who do not agree to participate in the study.
* Contraindication to central venous or arterial catheterization.
* Patients who were already treated in ICU because of sepsis or septic shock before this surgery.
* Known chronic renal failure.
* Re-laparotomy.
* Peritonitis due to acute mesenteric ischaemia, thrombosis or trauma.
* Dying patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2016-01; Primary Completion 2017-01-01 (Actual); Study Completion 2018-02-01 (Actual)

PRIMARY OUTCOMES:
Inpatient mortality in both treatment arms. | 30 days intra-hospital mortality
  Comparison of 30 days intra-hospital mortality in both arms.

SECONDARY OUTCOMES:
Comparison of incidence of severe hypotension MAP <65 mmHg after anaesthesia induction in both arms. | 1-5 minutes after anaesthesia induction.
  To evaluate the incidence of severe hypotension after anesthesia induction (1 - 5 minutes after induction) in both groups.
Comparison of fluid management in both arms (from hospitalisation to the surgery, during the surgery, after the surgery up to 24 hours). | up to 24 hours
  Comparison of tow fluids management strategies. Usual monitoring group - fluid management based on fluid responsiveness based by clinical sings. FATE group - fluid management based on focused transthoracic echocardiography data.
Comparison of septic shock incidence in both arms. | up to 30 days
  To compare the manifestation of septic shock (hemodynamics instability not responding to fluid administration, which requires norepinephrine infusion to maintain MAP ≥ 65 mmHg);
Number of ICU-Free days. | up to 30 days
  To compare ICU free days in both groups.

CONTACTS AND LOCATIONS:
Overall Officials: Andrius Macas, profesor, Study Chair — Lithuanian university of health sciencies
Locations (1):
- Lithuanian university of health sciencies, Kaunas, A. Mickeviciaus Street 9, Lithuania

IPD SHARING:
Plan to Share IPD: No